CLINICAL TRIAL: NCT01347190
Title: A Double Blind, Randomized, Placebo Controlled, Single Dose, Phase I Study of the Safety and Tolerability of Alpha1 Proteinase Inhibitor (Human) Inhalation Solution (CR002) in Subjects With Cystic Fibrosis
Brief Title: Safety and Tolerability Study of Liquid Alpha1 Proteinase Inhibitor (API) in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002_1004; 2010-022671-60 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Liquid API (Experimental)
  Interventions: Biological: CR002 Liquid API
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CR002 Liquid API — A single nominal dose of CR002 (three different dose groups) will be inhaled as an aerosol mist produced by an I-neb Adaptive Aerosol Delivery (AAD) System.
  Arms: Liquid API
Biological: Placebo — A single nominal dose of Placebo will be inhaled as an aerosol mist produced by an I-neb Adaptive Aerosol Delivery (AAD) System.
  Arms: Placebo

SUMMARY:
Study to assess safety and tolerability of a single dose of study-drug administered to Cystic Fibrosis (CF) patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of CF: one or more clinical findings consistent with CF and at least one of the following:

  1. Sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test OR
  2. A genotype with two identifiable mutations consistent with CF (∆F508 homozygous or two alleles known to cause a class I, II, or III mutation)
* Have an FEV1 ≥30% of predicted normal as defined by age, gender, and height

Exclusion Criteria:

* Oxygen saturation <90%
* Changed in treatment regimen within 2 weeks prior to screening
* Antibiotics regimen change < 4 weeks before screening
* Persistent colonization with Burkholderia cepacia
* Serum IgA < 50% of lower level of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse events | 44 Days (Day -21 to Day 22)

CONTACTS AND LOCATIONS:
Overall Officials: Program director Clinical R&D, Study Director — CSL Behring
Locations (11):
- Bulgaria (2):
  - Site 11, Sofia
  - Site 12, Varna
- Site 30, Debrecen, Hungary
- Poland (5):
  - Site 24, Bialystok
  - Site 22, Gdansk
  - Site 21, Poznan
  - Site 20, Rabka-Zdrój
  - Site 23, Warsaw
- United Kingdom (3):
  - Site 42, Papworth Hospital
  - Site 40, Penarth
  - Site 41, Southampton